CLINICAL TRIAL: NCT00626769
Title: Safety Profile and Bone Efficacy of the Phytoestrogen Genistein in a Cohort of Osteopenic, Postmenopausal Women After Three Years of Treatment: a Follow-up Study
Brief Title: Third Year Evaluation on Genistein Efficacy and Safety
Status: Completed | Type: Observational
Sponsor: University of Messina (Other)
Collaborators: Primus Pharmaceuticals (Industry)
Responsible Party: Prof. Francesco Squadrito, University of Messina
Other Study IDs: 2005-07
Record Dates: First submitted 2008-02-19; First posted 2008-02-29 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Menopause; Osteopenia
Keywords: Genistein; Bone mineral density; digital mammography; safety
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, urine.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Postmenopausal women with established osteopenia receiving aglycone genistein 54 mg/day for 3 years
  Interventions: Dietary Supplement: aglycone genistein
- 2: Postmenopausal women with established osteopenia receiving placebo (Calcium and vitD) for 3 years
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: aglycone genistein — 2 capsules per day containing 27 mg of aglycone genistein, calcium carbonate (500 mg) and vitamin D (400 IU), for a 3-year period.
  Other Names: Genivis; Fosteum
  Groups: 1
Dietary Supplement: placebo — 2 capsules per day containing calcium carbonate (500 mg) and vitamin D (400 IU), for a 3-year period.
  Groups: 2

SUMMARY:
BACKGROUND: Recent evidences showed that the phytoestrogen genistein positively affects bone metabolism with no clinically significant adverse effects in a cohort of osteopenic, postmenopausal women. However, there is still a knowledge gap regarding the long-term safety of genistein on the breast, the uterus, the thyroid gland and its efficacy in postmenopausal women.

OBJECTIVE: To assess the safety profile of genistein on mammary and thyroid glands and endometrium and cardiovascular apparatus and its effects on bone metabolism after a 3-year therapy with pure, standardized genistein (54 mg/day).

DETAILED DESCRIPTION:
DESIGN: The parent study was a randomized, double-blind, placebo-controlled trial involving 389 osteopenic, postmenopausal women for 24 months. After the 24-month visit, a sub-population (138 patients) accepted to continue the intervention until 36 months, thus generating a follow-up study.

SETTING: 3 Italian university medical centers. INTERVENTIONS: Participants received 54 mg of genistein, daily, (n=71) or placebo (n=67). Both intervention and placebo contained calcium and vitamin D3. All patients also received dietary instruction in an isocaloric fat-reduced diet.

MEASUREMENTS: Mammographic breast density at baseline and after 24 and 36 months was assessed by visual classification scale and by digitized quantification. BRCA1 and BRCA2 molecular message, sister chromatid exchanges and endometrial thickness were also evaluated at the same time points. Measurements of lumbar spine and femoral neck BMD and QUS t-score were assayed in our patients. Secondary outcomes were serum levels of B-ALP, IGF-I, sRANKL, osteoprotegerin and urinary excretion of CTX, pyridinoline and deoxypyridinoline. Furthermore insulin resistance (HOMA-IR), glucose levels, homocysteine and hot flushes were also evaluated. In addition for thyroid safety TSH, fT3, fT4, thyroid autoantibodies, and mRNA for thyroid and retinoid receptors were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Have not had a menstrual period in the preceding year
* Had not undergone surgically induced menopause
* Had a follicle-stimulating hormone level > 50 IU/liter and a serum 17 beta-estradiol level ≤ 100 pmol/liter
* Established osteopenia (-1<T-score<-2.5 SD)

Exclusion Criteria:

* Clinical or laboratory evidence of confounding systemic diseases, such as cardiovascular, hepatic, or renal disorders
* Coagulopathy, use of oral or transdermal estrogen, progestin, androgen or other steroids
* Biphosphonates, cholesterol-lowering therapy or cardiovascular medications in the preceding six months
* Smoking habit of more than two cigarettes per day
* Previous treatment with any drug that could affect the skeleton in the preceding year
* A family history of estrogen-dependent cancer
* BMD at femoral neck > 0.795 g/cm2; this BMD value corresponds to a T score of -1 standard deviation

Ages: 49 Years to 67 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women (age 49-67 yrs)
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2005-07; Primary Completion 2006-07 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | basal and after 1 year
Mammographic breast density | basal and after 3 years

SECONDARY OUTCOMES:
Bone-specific alkaline phosphatase (B-ALP) | basal and after 1 year
Insulin-like growth factor 1 (IGF-1) | basal and after 1 year
Pyridinium cross-links (pyridinoline and deoxypyridinoline) | basal and after 1 year
carboxy-terminal cross-linking telopeptide (CTX) | basal and after 1 year
Osteoprotegerin and soluble receptor activator of NF-kB ligand (s-RANKL) | basal and after 1 year
BRCA1 and BRCA2 mRNA levels | basal and after 3 years
Sister Chromatid exchanges | basal and after 3 years
Endometrial thickness | basal and after 3 years
Insulin resistance | basal and after 3 years
hot flushes | basal and after 3 years
Thyroid status | basal and after 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Squadrito, MD, Principal Investigator — University of Messina; Rosario D'Anna, MD, Study Director — University of Messina

REFERENCES:
- [Background] Marini H, Minutoli L, Polito F, Bitto A, Altavilla D, Atteritano M, Gaudio A, Mazzaferro S, Frisina A, Frisina N, Lubrano C, Bonaiuto M, D'Anna R, Cannata ML, Corrado F, Adamo EB, Wilson S, Squadrito F. Effects of the phytoestrogen genistein on bone metabolism in osteopenic postmenopausal women: a randomized trial. Ann Intern Med. 2007 Jun 19;146(12):839-47. doi: 10.7326/0003-4819-146-12-200706190-00005. PMID 17577003
- [Derived] Bitto A, Polito F, Atteritano M, Altavilla D, Mazzaferro S, Marini H, Adamo EB, D'Anna R, Granese R, Corrado F, Russo S, Minutoli L, Squadrito F. Genistein aglycone does not affect thyroid function: results from a three-year, randomized, double-blind, placebo-controlled trial. J Clin Endocrinol Metab. 2010 Jun;95(6):3067-72. doi: 10.1210/jc.2009-2779. Epub 2010 Mar 31. PMID 20357174
- [Derived] Marini H, Bitto A, Altavilla D, Burnett BP, Polito F, Di Stefano V, Minutoli L, Atteritano M, Levy RM, D'Anna R, Frisina N, Mazzaferro S, Cancellieri F, Cannata ML, Corrado F, Frisina A, Adamo V, Lubrano C, Sansotta C, Marini R, Adamo EB, Squadrito F. Breast safety and efficacy of genistein aglycone for postmenopausal bone loss: a follow-up study. J Clin Endocrinol Metab. 2008 Dec;93(12):4787-96. doi: 10.1210/jc.2008-1087. Epub 2008 Sep 16. PMID 18796517